CLINICAL TRIAL: NCT00983216
Title: A One-Directional, Open-Label Drug Interaction Study to Investigate the Effects of Multiple-Dose Ketoconazole on Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between Colchicine and Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1012
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: blood levels over time;; pharmacokinetics;; healthy adult;; cytochrome p450
MeSH Terms: interventions — Colchicine; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): -baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Steady-State Ketoconazole (Experimental): -colchicine pharmacokinetics in presence of steady-state ketoconazole
  Interventions: Drug: Ketoconazole; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of colchicine 0.6 mg administered alone at 7:30 a.m. on Day 1.
  Other Names: COLCRYS TM
  Arms: Colchicine alone
Drug: Ketoconazole — one 200 mg Ketoconazole tablet administered twice daily at 7:15 a.m. and 7:15 p.m. on Days 15-18 without regard to meals, then along with colchicine at 7:15 a.m. on Day 19 after an overnight fast of at least 10 hours; final dose of 200 mg administered at 7:15 p.m. on Day 19
  Arms: Colchicine with Steady-State Ketoconazole
Drug: Colchicine — A single dose of colchicine 0.6 mg administered along with ketoconazole at 7:15 a.m. on Day 19 after an overnight fast of at least 10 hours
  Arms: Colchicine with Steady-State Ketoconazole

SUMMARY:
Ketoconazole is a potent inhibitor of the cytochrome P450 (CYP) 3A4 enzyme system, one of the enzyme systems responsible for the metabolism of colchicine. This study will evaluate the effect of multiple doses of ketoconazole on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Ketoconazole is a potent inhibitor of the cytochrome P450 (CYP) 3A4 enzyme system, one of the enzyme systems responsible for the metabolism of colchicine. This study will evaluate the effect of multiple doses of ketoconazole on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period. After a fast of at least 10 hours, twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 years will be given one dose of colchicine (1 x 0.6 mg tablet) orally on Day 1. Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for twenty-four hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will then continue on a non-confined basis on Days 2-5. On Days 15-18, subjects will return to the clinic daily for non-confined dosing of ketoconazole (1 x 200 mg tablet) twice daily, every 12 hours. Administered ketoconazole doses on these days will not necessarily be in a fasted state. On Day 15, after taking the first dose of ketoconazole, subjects will remain in the clinic for observation for 1 hour post-dose administration. Then, on Day 19, co-administration of a single dose of colchicine (1 x 0.6 mg tablet) and ketoconazole (1 x 200 mg tablet) will occur following a fast of at least 10 hours in subjects confined to the clinic for dosing and 24-hour blood sampling will be performed at times sufficient to adequately determine the pharmacokinetics of colchicine. Blood sampling will continue on a non-confined basis on Days 20-23. Fasting will continue for 4 hours following the co-administered dose of ketoconazole and colchicine. The final dose of ketoconazole (1 x 200 mg tablet) will be administered to subjects the evening of Day 19, in a non-fasting state. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (blood pressure and pulse) will be measured prior to dosing and at 1, 2, and 3 hours following drug administration on Days 1 and 19 to coincide with peak plasma concentrations of both colchicine and ketoconazole. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff, will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine or ketoconazole or any other anti-fungal agent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS - Cetero
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, male and female volunteers, consisting of volunteers from the community at large, were enrolled in the study.
Pre-assignment Details: 55 subjects were screened, 12 were screen failures, 7 had schedule conflicts, 1 was not used due to history of non-compliance, and 12 were not needed
Groups:
- Colchicine Alone / With Ketoconazole (at Steady-state): [All subjects received each of the study treatments.] Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast, followed by a washout period of 14 days. On Day 15, subjects began taking one 200 mg ketoconazole tablet twice daily at 7:15 a.m. and at 7:15 p.m. without regard to meals. Then, on Day 19, each subject received both one 0.6 mg colchicine tablet and one ketoconazole 200 mg tablet at 7:15 a.m. after an overnight fast. A final dose of ketoconazole was administered at 7:15 p.m. that evening.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Ketoconazole (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone / With Ketoconazole (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0
Period: Ketoconazole Alone
Arm/Group | Colchicine Alone / With Ketoconazole (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0
Period: Colchicine With Ketoconazole
Arm/Group | Colchicine Alone / With Ketoconazole (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone / With Ketoconazole (at Steady-state)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — age range: ≥18 and ≤45 years
  Participants
    <=18 years | 2
    Between 18 and 65 years | 22
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn within 1 hour prior to colchicine dosing (0 hour) on Days 1 and 19, and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours after colchicine dose administration
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast, followed by a washout period of 14 days.
- Colchicine With Ketoconazole (at Steady-state): On Day 15, subjects began taking ketoconazole 200 mg twice daily at 7:15 a.m. and at 7:15 p.m. without regard to meals. Then, on the morning of Day 19 after an overnight fast of at least 10 hours, all subjects received a single dose of colchicine 0.6 mg along with ketoconazole 200 mg. A final dose of ketoconazole was administered at 7:15 p.m. that evening.
Arm/Group | Colchicine Alone | Colchicine With Ketoconazole (at Steady-state)
Number analyzed (Participants) | 24 | 24
pg/mL | 2,779.08 (1,036.89) | 5,266.92 (1,461.66)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the colchicine plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Ketoconazole (at Steady-state)
Number analyzed (Participants) | 24 | 24
pg-hr/mL | 11,988.61 (4,836.01) | 34,382.82 (9,445.74)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the colchicine plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Ketoconazole (at Steady-state)
Number analyzed (Participants) | 24 | 24
pg-hr/mL | 14,314.09 (5,991.79) | 43,680.90 (11,673.08)

ADVERSE EVENTS:
Groups:
- Ketoconazole Alone: On Day 15 to 18, subjects took ketoconazole 200 mg twice daily at 7:15 a.m. and at 7:15 p.m. without regard to meals.
- Colchicine With Ketoconazole (at Steady-state): On the morning of Day 19 after an overnight fast of at least 10 hours, all subjects received a single dose of colchicine 0.6 mg along with ketoconazole 200 mg. A final dose of ketoconazole was administered at 7:15 p.m. that evening.
Arm/Group | Colchicine Alone | Ketoconazole Alone | Colchicine With Ketoconazole (at Steady-state)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3 | 3 | 8
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Ketoconazole Alone | Colchicine With Ketoconazole (at Steady-state)
nausea (Gastrointestinal disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
dizziness (Nervous system disorders) | 0/24 (0) | 0/24 (0) | 2/24 (2)
headache (Nervous system disorders) | 3/24 (3) | 3/24 (4) | 5/24 (6)
polymenorrhoea (Reproductive system and breast disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days